CLINICAL TRIAL: NCT01717807
Title: C11-Erlotinib PET/CT as a Tool for Identification and Characterization of Tumor With High Expression of Epidermal Growth Factor Receptor(EGFR).
Acronym: EGFR; PET/CT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0365-12-HMO
Record Dates: First submitted 2012-10-28; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer; Pancreatic Cancer
Keywords: epithelial growth factor receptors; lung cancer; advanced tumor of pancrease; erlotinib; C11-Erlotinib PET/CT
MeSH Terms: conditions — Lung Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- lung cancer; advanced pancreatic cancer
  Interventions: Other: C11-Erlotinib PET/CT

INTERVENTIONS:
Other: C11-Erlotinib PET/CT

SUMMARY:
The EGFR is one of the most frequently overexpressed proteins in various cancers including lung cancer, and is related to tumor progression and resistance to most treatments.

New treatment strategies targeting EGFR have been developed: "although much work remains to be done, erlotinib has already established itself as part of the therapeutic armamentarium against cancer"(A review of erlotinib and its clinical use. Tang PA, Tsao MS, Moore MJ. Expert Opin Pharmacotherapy. 2006 Feb;7(2):177-93.)

Noninvasive PET/CT imaging of EGFR expression activity and mutation status in NSCLC could aid in the selection of patients for individualized therapy with EGFR kinase inhibitors.

Whole-body noninvasive PET/CT imaging could estimate treatment-responsive vs. -resistant tumor burden before the initiation of therapy with EGFR inhibitors.

The purposes of the study are:

1. To adjust an optimal treatment for patients with tumors that have high expression of EGFR by identification of this type of cancer using C11-Erlotinib PET/CT during pretreatment work-up; as well as to follow up after treatment response.
2. To recognize patients with advanced pancreatic cancer responding to treatment with erlotinib and to distinguish them from non-responders.

ELIGIBILITY:
Inclusion Criteria:

* patients with NSC type of lung cancer with high expression of EGFR who are candidates for erlotinib as second / third line of treatment;
* patients with advanced pancreatic tumor who are candidates for complex gemcitabine and erlotinib treatment.

Exclusion Criteria:

* lack of histological diagnosis;
* not a candidate for erlotinib;
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: oncological patients with NSC type of lung cancer and with advanced pacreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Measure of extent and intensity ( by standardized uptake value - SUV) of C11-Erlotinib accumulation by tumors and metastasis before and after treatment

SECONDARY OUTCOMES:
size of tumor and metastasis (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel